CLINICAL TRIAL: NCT01989533
Title: Phase I Study of Safety and Immunogenicity of Ad4-HIV Vaccine Vectors in Healthy Volunteers
Brief Title: Study of Safety and Immunogenicity of HIV Vaccines in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 140011; 14-I-0011
Record Dates: First submitted 2013-11-19; First posted 2013-11-21 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-04-24

CONDITIONS: Vaccine Response
Keywords: HIV Vaccine; Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- A (Placebo Comparator): Placebo controlled (blinded)
  Interventions: Biological: Ad4-mgag; Biological: Ad4-EnvC150; Biological: gp 120 Protein Boost
- B (Active Comparator): Intranasal Randomized
  Interventions: Biological: Ad4-mgag; Biological: Ad4-EnvC150; Biological: gp 120 Protein Boost
- C (Experimental): Oral Open label
  Interventions: Biological: Ad4-mgag; Biological: Ad4-EnvC150; Biological: gp 120 Protein Boost
- D (Experimental): Intranasal Open Label
  Interventions: Biological: Ad4-mgag; Biological: Ad4-EnvC150; Biological: gp 120 Protein Boost

INTERVENTIONS:
Biological: Ad4-mgag — Ad4 live virus vaccine with an HIV insert
Biological: Ad4-EnvC150 — Ad4 live virus vaccine with an HIV insert
Biological: gp 120 Protein Boost — HIV protein boost

SUMMARY:
Background:

- Vaccines create resistance to disease. This study tests experimental human immunodeficiency virus (HIV) vaccines that use an adenovirus as a transporter. Transporters may help vaccines stimulate an immune response against HIV. This means the body works to fight infection. Researchers want to see if different ways of giving the vaccines cause different immune responses. They also want to see if the vaccines adenovirus is contagious. Adenoviruses cause cold symptoms or mild eye infections.

Participants cannot get HIV from these vaccines. But they can get the adenovirus, so their entire household and intimate contacts must participate.

Objective:

- To test the safety of experimental HIV vaccines.

Eligibility:

- Healthy adults 18-49 years old.

Design:

* Participants will be screened with medical history, physical exam, and blood and urine tests.
* Participants will receive the vaccine 3 times over 6 months. Each time, they will have a physical exam and blood and urine tests. Samples will be taken from their nose, rectum, and cervix.
* Some participants will receive the vaccine by swallowing 11 capsules with water. Clinic staff will observe them for 1 hour.
* Some participants will receive the vaccine swabbed in their throat. They will get dose 1 at the hospital and stay there for 1 week. They will have medical tests and nose swabs. Doses 2 and 3 will not require a hospital stay.
* Participants will have 7 follow-up visits over 6 months, with a physical exam and blood tests. Samples will be taken from their nose, throat, and rectum.
* Household and intimate contacts will have 4 clinic visits over 8 months, with a physical exam and blood tests.

DETAILED DESCRIPTION:
This is a Phase 1, single center, randomized, double-blind study designed to evaluate the safety and immunogenicity of live, replication-competent recombinant Adenovirus type 4-HIV vaccine regimens. The oral route will also contain a placebo control. The vaccine candidates Ad4-mgag and Ad4-EnvC150 will be formulated as enteric-coated capsules to be delivered orally, and as an aqueous formulation for intranasal administration. Determining the optimal regimen and route will greatly accelerate investigations of these vectors as HIV vaccine platforms.

Participants volunteering to receive the vaccine orally will be randomized to 1 of 4 treatment arms, and those volunteering to receive the vaccine via the intranasal route will be randomized to 1 of 3 treatment arms. Participants will receive either 1 or both vaccines or placebo, depending on group assignment. The study vaccines will be administered to participants in 3 rounds of vaccination at 0, 2, and 6 months. All participants will receive a booster vaccination with a bivalent HIV gp120 glycoprotein at 8 months. Intranasal vaccine recipients with household contact(s) will receive the first vaccine in the NIH Special Clinical Studies Unit or other appropriate unit and be followed on an inpatient basis to allow for respiratory isolation. Intranasal vaccinees without household contact(s) may also receive the vaccination as inpatients or may opt to receive the vaccine on an outpatient basis if they agree to follow precautions for preventing the spread of adenovirus. Beginning 4 days after vaccination, inpatient participants will be tested daily for respiratory shedding of Ad4 by nasopharyngeal wash. They will be discharged to home with close monitoring on Day 7 or after 2 consecutive negative washes, whichever comes first; they may remain on the unit longer if medically necessary. Prior to receiving the second dose of vaccine on an outpatient basis, seroconversion to Ad4 will be confirmed in the intranasal vaccine recipients. Those who have household contact(s) and have not seroconverted will continue to receive subsequent doses as inpatients until they show seroconversion. Those who do not have household contact(s) and those who have seroconverted may receive the remaining vaccinations as inpatients or may opt to receive the doses on an outpatient basis if they agree to follow precautions for preventing the spread of adenovirus. If they decline these options, they may withdraw from the study and will be replaced. Oral capsule recipients will be vaccinated and discharged to home.

In addition to clinical and laboratory monitoring of safety, the principal assessments will be shedding of this viruses in rectal, cervicovaginal, throat, and nasal swabs, and assessment of the antibody (mucosal and systemic) response to the HIV and to the Ad4 virus.

The candidate vaccines will also be administered to 2 groups of participants who have previously received an unrelated HIV vaccine in another clinical study and/or are Ad4 seropositive. The aim for these groups is to explore the boost potential of the enteric coated capsule and aqueous formulations of the Ad4-mgag and Ad4- EnvC150 vaccines when given to subjects who have previously received another HIV vaccine and/or are Ad4 seropositive.

The adenovirus vaccines will not be retested for stability in 2018, and therefore will be out of specifications on May 9th 2018. In an effort to capture as much information on immunogenicity and adenoviral replication as possible, we will implemement the following change beginning in 2018. The study will continue with enrollment into the remaining treatment groups in a nonrandomized manner such that remaining participants receive both the Ad4-mgag and Ad4-EnvC150 intranasally. These participants will receive 2 rounds of the intranasal vaccine at Months 0 and 2 followed by a single dose of the booster vaccination at Month 4.

All participants will be followed for a total of 6 months following the final dose of study vaccine. Household and intimate contacts will also be enrolled and monitored for Adenovirus and HIV antibodies for up to 8 months.

ELIGIBILITY:
* INCLUSION CRITERIA:

All participants (vaccinees, household contacts, and intimate contacts) must meet all of the following criteria:

1. Age 18 to 49 years for vaccinees. Age 18 to 65 years for household and intimate contacts.
2. Negative FDA-approved HIV test.
3. Able to provide proof of identity to the acceptance of the Principal Investigator or designee during enrollment.
4. Available and willing to participate in follow-up visits and tests for the duration of the study.
5. Willing to have samples stored for future research.

The following inclusion criteria apply to vaccinees and intimate contacts, but not to household contacts:

1. In good general health without clinically significant medical history.
2. Willing to discuss HIV infection risks with the study clinicians, assessed as low risk for HIV infection, amenable to HIV risk reduction counseling, and committed to maintaining behavior consistent with

   low risk of HIV exposure through the last required clinic visit in the protocol schedule.
3. Negative Beta-HCG pregnancy test for females presumed to be of reproductive potential.
4. A female must meet one of the following criteria:

   1. No reproductive potential because of menopause (one year without menses) or because of a hysterectomy, bilateral oophorectomy, or tubal ligation.

      OR
   2. Participant agrees to be heterosexually inactive or consistently practice contraception at least 21 days prior to and 28 days following each vaccination. Acceptable methods of contraception include the following:

      * condoms, male or female, with a spermicide.
      * diaphragm or cervical cap with spermicide.
      * contraceptive pills, Norplant, or Depo-Provera.
      * male partner has previously undergone a vasectomy for which there is documentation.
      * intrauterine device.
5. Male participants must agree to practice abstinence or effective birth control for at least 21 days prior to and 28 days following each vaccination.

The following inclusion criteria apply only to vaccinees and not to household or intimate contacts:

1. Willing to receive HIV test results and abide by NIH guidelines for partner notification of positive HIV results.
2. Physical examination and laboratory results without clinically significant findings within the 8 weeks prior to enrollment.
3. Willing to avoid vaccination other than the study agent for 30 days prior to and 30 days after administration of the Ad4-HIV vaccine.
4. Safety Laboratory Criteria within 8 weeks prior to enrollment:

   Hematopoietic: -White blood cell count and Lymphocyte count +/- 25% of normal limits for the NIH Clinical Center
   * Platelet count of least 100,000/mm(3)
   * Hemoglobin >11.2 g/dL for females and >13.0 g/dL for males.

   Renal: BUN <23 mg/dL; creatinine within normal limits for the NIH Clinical Center

   Hepatic: Serum total bilirubin less than or equal to 2 mg/dL

   Metabolic: ALT <2 times upper limit of normal range

   Endocrine: Serum glucose within normal range
5. Additional Laboratory Criteria:

Immunologic: No history of hypogammaglobulinemia

Serologic: Ad4 neutralizing antibody 80% inhibitory dilution <1:100 (This criterion does not apply to participants in Arms C and D.)

The following inclusion criterion applies only to intranasal vaccinees and not to capsule vaccine recipients or household or intimate contacts:

1. Willing to either:

1. be hospitalized at the Clinical Center under respiratory precautions for up to 7 days or longer if medically indicated (required for those with household contact(s) until they show seroconversion); or
2. follow precautions for preventing the spread of adenovirus in the community.

EXCLUSION CRITERIA:

A participant (vaccinees, household contacts, and intimate contacts) will be excluded if they have the following:

1. Any condition that, in the investigator s judgement, places the subject at undue risk by participating in the study.

The following exclusion criterion applies to vaccinees and intimate contacts, but not to household contacts:

1. History of any prior disease or therapy which would affect immune or pulmonary function.
2. Prior malignancy, except curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
3. History of radiation therapy or cytotoxic/cancer chemotherapy.
4. History of diabetes mellitus.
5. Immunodeficiency or autoimmune disease.
6. Acute infection or a recent (within 6 months) history of chronic infection suggestive of immunodeficiency.
7. Taking any medication which may affect immune function, except participants may be taking low doses of nonprescription strength NSAIDS (including e.g. ibuprofen or aspirin) or acetaminophen.
8. Chronic respiratory disorders including asthma, emphysema, interstitial lung disease, pulmonary hypertension, recurrent pneumonia, or recent or ongoing respiratory tract infection. If a respiratory disorder is transient, defer immunization but do not exclude the participant.
9. Active Hepatitis B or C infection (i.e. Hepatitis B or C positive serology with the presence of virus antigen or DNA. Ongoing viral replication will be confirmed by a Hepatitis B antigen or Hepatitis C viral load).
10. Female of child-bearing potential who is breast-feeding or planning pregnancy during the 28 days following vaccination.

The following exclusion criteria apply only to vaccinees and not to household or intimate contacts:

1. Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgment of the investigator, would interfere with or serve as a contraindication to receipt of live virus vaccine, protocol adherence, or a participant s ability to give informed consent.
2. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years; disorder requiring lithium; or suicidal ideation occurring within five years prior to enrollment.
3. Participants that live in the same house or apartment with any of the following will be excluded:

   1. An individual under 18 years of age.
   2. An elderly individual (>65 years of age).
   3. An immunocompromised or immunosuppressed individual.
   4. An individual with chronic respiratory disease.
   5. A woman who is currently pregnant or planning a pregnancy during the period of immunization.
4. Healthcare worker who has direct contact with immunodeficient, unstable patients, or pediatric patients.
5. Participants caring for children <18 years of age.
6. Receipt of any of the following:

   * Antiviral medications within 30 days prior to vaccination.
   * Blood products within 120 days prior to HIV screening.
   * Immunoglobulin within 60 days prior to HIV screening.
   * Investigational research drugs or any other investigational agent that in the judgement of the Principal Investigator might interact with the study vaccine within 30 days prior to initial study vaccine administration.
   * Allergy treatment with antigen injections within 30 days of study vaccine administration.
7. History of Guillain-Barr(SqrRoot)(Copyright) syndrome.
8. Indeterminate HIV Western Blot test.
9. Prior receipt of an Ad5-based vaccine.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2013-11-19; Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of the Ad4-mgag and Ad4-EnvC150 vaccines in humans when administered via the oral or intranasal route. | Ongoing
  Safety

SECONDARY OUTCOMES:
To evaluate the immunogenicity of the Ad4- mgag and Ad4-EnvC150 vaccines in humans when administered via the oral or intranasal routes in humans | Ongoing
  Immunogenicity response

CONTACTS AND LOCATIONS:
Overall Officials: Mark Connors, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Boyaka PN, Tafaro A, Fischer R, Leppla SH, Fujihashi K, McGhee JR. Effective mucosal immunity to anthrax: neutralizing antibodies and Th cell responses following nasal immunization with protective antigen. J Immunol. 2003 Jun 1;170(11):5636-43. doi: 10.4049/jimmunol.170.11.5636. PMID 12759444
- [Background] Brandt CD, Kim HW, Vargosko AJ, Jeffries BC, Arrobio JO, Rindge B, Parrott RH, Chanock RM. Infections in 18,000 infants and children in a controlled study of respiratory tract disease. I. Adenovirus pathogenicity in relation to serologic type and illness syndrome. Am J Epidemiol. 1969 Dec;90(6):484-500. doi: 10.1093/oxfordjournals.aje.a121094. No abstract available. PMID 4312064
- [Background] Braucher DR, Henningson JN, Loving CL, Vincent AL, Kim E, Steitz J, Gambotto AA, Kehrli ME Jr. Intranasal vaccination with replication-defective adenovirus type 5 encoding influenza virus hemagglutinin elicits protective immunity to homologous challenge and partial protection to heterologous challenge in pigs. Clin Vaccine Immunol. 2012 Nov;19(11):1722-9. doi: 10.1128/CVI.00315-12. Epub 2012 Aug 29. PMID 22933397